CLINICAL TRIAL: NCT05789446
Title: Confirmatory Efficacy of the Building a Strong Identity and Coping Skills Program for Low-income and Minoritized Young Adolescents
Brief Title: Confirmatory Efficacy of the Building a Strong Identity and Coping Skills Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Martha E. Wadsworth, Professor of Psychology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAR-21-132
Record Dates: First submitted 2023-02-09; First posted 2023-03-29 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Stress; Anxiety; Depression
Keywords: Poverty; Discrimination; Stress; Coping
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BaSICS Intervention (Experimental): Intervention = Building a String Identity and Coping Skills (BaSICS). Children randomized to participate in 16 twice weekly BaSICS intervention sessions. Children learn coping skills, identity development, and collective action as ways to buffer against chronic stress.
  These children also complete pre- and post-intervention assessments, as well as 6-month and 12-month follow-up assessments.
  Interventions: Behavioral: Building a Strong Identity and Coping Skills
- Control (No Intervention): These children complete assessments only--timed to coincide with the intervention groups' assessments: pre- and post-intervention assessments, as well as 6-month and 12-month follow-up assessments. No intervention.

INTERVENTIONS:
Behavioral: Building a Strong Identity and Coping Skills — Psychoeducational program to teach children coping skills, healthy identity development, and collective social action
  Other Names: BaSICS
  Arms: BaSICS Intervention

SUMMARY:
The goal of this clinical trial is to the efficacy of the Building a Strong Identity and Coping Skills intervention within a sample of low-income and minoritized youth aged 11-14 who are seeking mental health treatment and have been placed on a waitlist to receive services.

The aims of this study are to: (1) confirm the efficacy of BaSICS by replicating previous findings, (2) Examine the changes of coping mechanisms and symptom change over the course of the BaSICS intervention, and (3) test models of physiologic stress reactivity and regulation to capture biological "risk" and recalibration.

Cohorts of 20 participants will randomly be enrolled in either the intervention (10) or control (10) groups. Participants enrolled in the intervention group will complete the BaSICS program and participants enrolled in the no intervention group will not be enrolled in the intervention program. The BaSICS program is designed to help treat anxiety, depression, and post-traumatic stress symptoms and disorders and have direct effects on physiologic stress response systems (hypothalamic-pituitary-adrenal (HPA) axis). Researchers will compare the intervention and no intervention groups to see if there is a difference in the reduction of markers for anxiety, depression, and suicide scores, changes in coping mechanism, and HPA reactivity profiles

ELIGIBILITY:
Inclusion Criteria:

* Children ages 11-14 at intake
* Family income at or below 200% federal poverty level
* Child speaks English
* Parent speaks English or Spanish

Exclusion Criteria:

* Intellectual disability
* Autism spectrum disorder
* High suicidal risk (score of 17 or more on the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-Kid))
* Severe depression (score of 19 or more on Patient health questionnaire (PHQ).

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Pre-post (3 months) and Pre-follow up (6 and 12 months)
  Changes in the number of anxiety problems that children report. Anxiety problems will be measured using the Screen for Child Anxiety Related Disorders (SCARED), Child Behavior Checklist (CBCL), and Youth Self Report (YSR).
Depression | Pre-post (3 months) and Pre-follow up (6 and 12 months)
  Changes in the number of depressive symptoms that children report. Depressive symptoms will be measured using the Patient Health Questionnaire (PHQ-9A), CBCL, and YSR.
Suicide Risk Markers | Pre-post (3 months) and Pre-follow up (6 and 12 months)
  Changes in the number of suicide risk markers that children report. Suicide risk markers will be measured using the Child Trauma Screen (CTS) and Mini Kid.

SECONDARY OUTCOMES:
Engagement Coping Skills Acquisition | Pre-post (3 months) and Pre-follow up (6 and 12 months)
  Changes in the number of coping skills that children can report. Engagement Coping Skills Acquisition will be assessed with the Responses to Stress Questionnaire (RSQ), Children's Sadness Management Scale (CSMS) and Coping Skills Scale (CSS).
HPA Reactivity Profile | Pre-post (3 months) and Pre-follow up (6 and 12 months)
  Changes in levels of salivary cortisol across a 90-minute Trier Social Stress Test (TSST) protocol
Collaborative Coping | Pre-post (3 months) and Pre-follow up (6 and 12 months)
  Changes in the number of collaborative coping skills that children report. Collaborative Coping will be assessed with the Collaborative Coping Discussion, Youth Civic and Character Measure (YCCM), and Social Skills Improvement System (SSIS).
Sociocultural Identity Development | Pre-post (3 months) and Pre-follow up (6 and 12 months)
  Changes in the sociocultural identity beliefs that children report. Sociocultural identity beliefs will be assessed with the Child and Adolescent Social Support (CASS), Early Identity Exploration Scale (EIES), and Multigroup Ethnic Identity Measure (MEIM).

CONTACTS AND LOCATIONS:
Overall Officials: Martha E Wadsworth, PhD, Principal Investigator — Penn State University
Locations (5):
- United States (5):
  - Pennsylvania Psychiatric Institute, Harrisburg, Pennsylvania
  - Penn State Health Medical Group - Psychiatry and Behavioral Health, Hershey, Pennsylvania
  - Penns Valley Area School District, Spring Mills, Pennsylvania
  - Dr. Edwin L. Herr Clinic, State College, Pennsylvania
  - Penn State Psychological Clinic, State College, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All data produced in the course of the project will be preserved and shared after de-identification. Item level spreadsheet data for all variables will be shared openly once cleaned. Data will be deposited into the National Institute of Mental Health Data Archive.
Time Frame: Data will become available after de-identification and cleaning.